CLINICAL TRIAL: NCT00130520
Title: Phase II Open-Label Trial of Erlotinib (Tarceva) and Bevacizumab in Women With Advanced Ovarian Cancer
Brief Title: Bevacizumab and Erlotinib Study in Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC #05-47;AVF3117s; NCT00696670 (obsolete NCT alias)
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Results first posted 2010-12-14 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2010-12

CONDITIONS: Ovarian Neoplasms
Keywords: advanced ovarian cancer; refractory ovarian cancer; primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label (Experimental)
  Interventions: Drug: bevacizumab; Drug: erlotinib

INTERVENTIONS:
Drug: bevacizumab — 10mg/kg every two weeks IV-bevacizumab
  Other Names: Avastin
Drug: erlotinib — 150mg daily by mouth-erlotinib
  Other Names: Tarceva

SUMMARY:
The purpose of this project is to determine if a new combination of drugs, erlotinib (Tarceva™) and bevacizumab is safe and effective for treating women diagnosed with ovarian cancer whose cancer has progressed while on prior standard chemotherapy treatment with a taxane (paclitaxel or docetaxel) and a platinum (cisplatin or carboplatin).

DETAILED DESCRIPTION:
Erlotinib and bevacizumab, novel biologics, offer a new regimen for the treatment of ovarian cancer in women who are refractory to standard drug regimens. Because bevacizumab is an anti-angiogenesis drug and erlotinib is an EGFR receptor inhibitor their combination would lead to the inhibition of multiple signal transduction pathways and the reversal of cancer progression in this difficult to treat population. The study seeks to determine the efficacy and safety of the EGFR receptor inhibitor, erlotinib plus the anti-angiogenesis VEGF ligand inhibitor bevacizumab in women with platinum and taxane refractory ovarian cancer.

The study design is a non-randomized, open label, single center Phase II trial using a Simon two stage design. Eligible patients are women who have a histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary or primary peritoneal carcinoma who have relapsed or are refractory to therapy after primary treatment of their disease.

Patients will be treated with erlotinib 150 mg/day orally and bevacizumab 10mg/kg every two weeks plus or minus one day intravenously. Forty patients will be enrolled in the study. Initially 20 eligible patients will be accrued. If one or no confirmed response is observed, the trial will be closed and the agents considered inactive. Otherwise, 20 additional eligible patients will be accrued for a total of 40 patients. Eight or more responses out of 40 will be considered evidence warranting further study of the agents provided other factors, such as progression-free and overall survival, also appear favorable.

Previous studies of this combination in non-small cell lung cancer, renal cell carcinoma and metastatic breast cancer have indicated a potential synergistic effect for these two agents. Preliminary data for the use of bevacizumab in advanced ovarian cancer indicates that this agent has single-agent activity. As a result, the researchers are interested in exploring the role of the combination of erlotinib and bevacizumab in advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary or primary peritoneal carcinoma.
* Relapsed after prior therapy with taxane and platinum-based therapy, within 6 months of completing, or had a best response of stable disease during no more than two prior chemotherapy treatments with a platinum (either cisplatin or carboplatin) and a taxane (paclitaxel or docetaxel). These agents may have been administered concurrently or sequentially. Besides the primary chemotherapy, two additional chemotherapy regimens are allowed. Hormonal therapy is allowed and will not be counted as a chemotherapy regimen.
* Up to one year of consolidation treatment with intraperitoneal and intravenous administered chemotherapy drugs to consolidate a clinical complete remission is allowed.
* Patients must have elevated CA-125 or measurable disease.
* For patients who do not have RECIST measurable disease, an elevated CA-125 (greater than two times the institutional upper limit of normal) will be required for enrollment.
* Debulking surgery for relapsed disease is allowed but must be completed at least 28 days prior to the first day of study therapy. Patient must have recovered from all side effects of surgery including a completely healed surgical incision.
* Patient must have a Zubrod performance status of 0-1.
* Patient must have adequate hepatic function as defined by:

  * a serum bilirubin ≤1.5 x the institutional upper limit of normal (IULN),
  * SGOT or SGPT ≤2.5 x the institutional upper limit of normal obtained within 14 days prior to start of therapy
* Patient must have an adequate renal function as defined by:

  * a serum creatinine ≤1.5 x the institutional upper limit of normal obtained within 14 days prior to start of therapy and a urine protein:creatinine (UPC) ratio of ≤ 1.0.
* Patients must be able to take oral medications
* Patients may not have ongoing problems with bowel obstruction or short bowel syndrome characterized by grade 2 or greater diarrhea or malabsorptive disorders.
* Patients must have the following hematological criteria:

  * Hemoglobin of >10gm/dL,
  * White blood cell count >2500,
  * Platelets >80,000
* Patients must be ≥ 18 years of age.

Exclusion Criteria:

* Subjects with mixed mullerian tumors and borderline ovarian tumors are excluded. Patients with a history of borderline ovarian tumors that have evolved into higher grade tumors will be eligible.
* The patient must not have received chemotherapy, biologic therapy or any other investigational drug for any reason within 28 days prior to start of therapy and must have recovered from toxicities of prior therapy to grade 1 or less with the exception of alopecia.
* Patient must not be pregnant or nursing because bevacizumab or erlotinib maybe harmful to the developing fetus and newborn. Women of reproductive potential must have a negative serum pregnancy test within 7 days prior to study consent. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
* Patients should not have psychological, familial, sociological, or geographical conditions that do not permit medical follow-up or compliance with the study protocol.
* Except for cancer-related abnormalities, patients should not have unstable or preexisting major medical conditions.
* Patients should not have any medical life-threatening complications of their malignancies
* Patients should not have a known severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, active uncontrolled infection, or HIV)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Baseline blood pressure of < or equal to 150/100 mmHg. Patients with a blood pressure reading above this level should be initiated on anti-hypertensive therapy and may be considered for protocol treatment when their blood pressure is adequately controlled.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction, cerebrovascular accident, transient ischemic attack, or unstable angina within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein:creatinine ratio > equal to 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
* Serious, non-healing wound, ulcer, or bone fracture
* Diagnosis of any other malignancy except non-melanomatous skin cancer in the past 5 years.
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Alberts, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Background] Chambers SK, Clouser MC, Baker AF, Roe DJ, Cui H, Brewer MA, Hatch KD, Gordon MS, Janicek MF, Isaacs JD, Gordon AN, Nagle RB, Wright HM, Cohen JL, Alberts DS. Overexpression of tumor vascular endothelial growth factor A may portend an increased likelihood of progression in a phase II trial of bevacizumab and erlotinib in resistant ovarian cancer. Clin Cancer Res. 2010 Nov 1;16(21):5320-8. doi: 10.1158/1078-0432.CCR-10-0974. PMID 21041183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting in June of 2005 and ended recruitment in January of 2008. All subjects were seen and treated at the Arizona Cancer Center in Tucson, Arizona.
Pre-assignment Details: The study had no pre-assignment criteria. This was an open label study and all subjects were given the same treatment.
Groups:
- Bevacizumab and Erlotinib: This is an open label study. All subjects received erlotinib 150 mg/day orally and bevacizumab 10 mg/kg intravenously every 2 weeks until disease progression. Progression free survival (PFS) was defined as the time from the start of therapy to the time of the first documentation of progression, symptomatic deterioration, or death due to any cause
Period: Overall Study
Arm/Group | Bevacizumab and Erlotinib
Started | 40 (85 women were screened for eligibility, 56 consented, 40 treated.)
Completion of at Least One Cycle | 39
Completed | 1
Not Completed | 39
Not completed — Adverse Event | 11
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 23
Not completed — Protocol non-compliance | 1
Not completed — Did not meet re-treatment criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Erlotinib
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 59.35 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Partial, Stable and Progression)
Description: Objective response was defined using standard RECIST criteria. CR(complete response)= disappearance of all target lesions PR(partial response)=30% decrease in the sum of the longest diameter of target lesions PD(progressive disease)=20% increase in the sum of the longest diameter of target lesions SD(stable disease)= small changes that do not meet above criteria
Time Frame: 06.16.2005 to 10.05.2009
Population: Population=subjects receiving 1 dose of intervention and one assessment post-baseline. One subject=not evaluable. Analysis-Enroll 40, initial accrual of 20. If ≤1 confirmed responses observed in 20=closure. If ≥2 responses=20 additional.
Measure: Number; unit: Participants
Arm/Group | Bevacizumab and Erlotinib
Number analyzed (Participants) | 39
Participants
  Complete Response | 1
  Partial Response | 8
  Stable Disease | 10
  Disease Progression | 20

2. Secondary Outcome: Progression Free Survival(PFS)
Description: PFS was defined as the time from the start of therapy to the time of the first documentation of progression(progression=20% increase in sum of longest diameters of target measurable lesions over smallest sum observed or baseline, progression of non-measurable disease in the opinion of treating physician, appearance of new lesion/site, Death due to disease), symptomatic deterioration (global deterioration of health status requiring discontinuation of treatment without objective evidence of progression), or death due to any cause;
Time Frame: June 2005 to October 5, 2009
Population: The population analyzed included all participants receiving at least 1 dose of study intervention and at least one assessment post-baseline. One subject was not evaluable. Analysis was per protocol
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab and Erlotinib
Number analyzed (Participants) | 39
months | 4 [1 to 26.8]

3. Primary Outcome: Median Response Duration (Weeks)
Description: Response duration=time (in weeks) between date of measurable response and date of progression (progression=20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed or baseline, progression of non-measurable disease in opinion of treating physician, any new lesion/site, death due to disease)if known or the date the subject went off protocol if they were still considered responders (ie do not qualify as progression) or are stable (Does not qualify for CR, PR, progression or Symptomatic Deterioration)
Time Frame: 1 week to 96 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: weeks
Arm/Group | Bevacizumab and Erlotinib
Number analyzed (Participants) | 39
weeks
  Responders | 36.1 [5.6 to 83.0]
  Stable | 25.6 [6.0 to 65.]

ADVERSE EVENTS:
Time Frame: Collected from the start of the 1st subject 6/2005 until the last subject was off treatment which was October 5, 2009 as the data was truncated for the purpose of the publication. Subjects came in for treatment every 2 weeks.
Arm/Group | Bevacizumab and Erlotinib
Serious Adverse Events (participants affected / at risk) | 12/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Erlotinib (N=40)
Hospitalization for dyspnea and fatigue (General disorders) | 1 (16)
hospitalization for diarrhea, nausea, vomiting and facial rash (CTCAE grade 2) (General disorders) | 1 (16)
Hospitalization for partial bowel obstruction (Gastrointestinal disorders) | 1 (16)
Hospitalizaton for diarrhea, abdomianl bloating, dyspnea (General disorders) | 1 (16) — Diagnosed as right pleural effusion
Death (General disorders) | 1 (16) — Death was due to disease progression and not study related
Myocardial infarct (Cardiac disorders) | 1 (16)
Bowel perforation-large intestine (Gastrointestinal disorders) | 1 (16)
Possible Myocardial infarction (Cardiac disorders) | 1 (16) — This MI was never confirmed and the investigator does not believe it was actually and MI
Abdominal fistula (Cardiac disorders) | 1 (16)
Nasal septal perforation (General disorders) | 1 (16)
Hospitalization for intercranial bleed (General disorders) | 1 (16) — This was never able to be confirmed
Hospitalization for fever (General disorders) | 1 (16)
Hospitilization for skin rash and pain (General disorders) | 1 (16)
Hospitilization for weakness and low hemoglobin (General disorders) | 1 (16)
Hospitalization for fatigue, dyspnea, weakness (General disorders) | 1 (16)
Hospitalization for headache and parasthesis (General disorders) | 1 (16)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and Erlotinib (N=40)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 7 (7)
Allergy/Immunology-Other (Immune system disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5) — Hemoglobin values out of normal range
Neutrophils/granuloctyes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (4) — Neutrophils/granulocytes out of normal range
Platelets (Blood and lymphatic system disorders) | 2 (2) — Platelet count out of normal range
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2)
Hypertension (Cardiac disorders) | 10 (10)
Constitutional Symptoms (Other) (General disorders) | 2 (2)
Fatigue (General disorders) | 16 (16)
Insomnia (General disorders) | 5 (5)
Rigors/chills (General disorders) | 3 (3)
Weight loss (General disorders) | 10 (10)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 13 (13)
Fever (in the absence of neutropenia) (General disorders) | 3 (3) — Neutropenia is defined as ANC<1.0x10e9/L
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4)
Nail Changes (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritius/itching (Skin and subcutaneous tissue disorders) | 6 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (9)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 31 (31)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 15 (15)
Dry Skin (Skin and subcutaneous tissue disorders) | 18 (18)
Constipation (Gastrointestinal disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 33 (33)
Distension/bloating, abdominal (Gastrointestinal disorders) | 8 (8)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dysphagia (difficulty swllowing) (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 5 (5)
Gastrointestinal-Other (Gastrointestinal disorders) | 12 (12)
Heartburn/dyspepsia (Gastrointestinal disorders) | 7 (7)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (clincal exam) (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 16 (16)
Taste alteration dysgeusia) (Gastrointestinal disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 14 (14)
Hemorrhage, GI (Gastrointestinal disorders) | 7 (7)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hemorrhage/Bleeding-Other (Blood and lymphatic system disorders) | 3 (3)
Infection (Infections and infestations) | 11 (11)
Infection (documented clinically or microbiologically) (Infections and infestations) | 5 (5) — with Grade 3 or 4 neutrophils (ANC<1.0x10e)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 5 (5)
Infection with unknown ANC (Infections and infestations) | 7 (7)
Edema:limb (Blood and lymphatic system disorders) | 3 (3)
Lymphatics-Other (Blood and lymphatic system disorders) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 27 (27)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 6 (6) — Out of normal laboratory range
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6 (6) — Outside of normal laboratory range
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 7 (7)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Proteinuria (Metabolism and nutrition disorders) | 5 (5)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 9 (9)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 10 (10)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 6 (6)
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 8 (8)
Ataxia (incoordination) (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 7 (7)
Mood Alteration (Psychiatric disorders) | 5 (5)
Neuropathy: cranial or sensory (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 2 (2)
Dry Eye Syndrome (Eye disorders) | 5 (5)
Ocular/Visual-Other (Eye disorders) | 4 (4)
Blurred Vision (Eye disorders) | 4 (4)
Pain (General disorders) | 21 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Renal/Genitourinary-other (Renal and urinary disorders) | 6 (6)
Urinary Frequency/Urgency (Renal and urinary disorders) | 2 (2)
Vaginal mucositis (Reproductive system and breast disorders) | 2 (2)
Vascular-Other (Vascular disorders) | 3 (3)
Pain-Other (General disorders) | 9 (9)
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No